CLINICAL TRIAL: NCT05373602
Title: The Incidence and Risk Factors of Low Anterior Resection Syndrome: Basing on Data of Chinese Patients From a Single Center
Brief Title: LARS for Chinese Patients
Status: Completed | Type: Observational
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Hongbo Wei, Vice-president of Third Affiliated Hospital, Sun Yat-Sen University, Third Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: LARS001
Record Dates: First submitted 2022-05-10; First posted 2022-05-13 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Incidence and Risk Factors of Low Anterior Resection Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: LARS questionnaire — Eligible participants were issued with LARS questionnaire (Chinese version) by E-mail, message, phone or face to face interview.

SUMMARY:
Low anterior resection syndrome (LARS) frequently occurs in patients undergoing low anterior resection (LAR). However, the incidence, exact mechanism and risk factors of major LARS largely variate in different studies. Considering varieties and differences of patient characteristics between Chinese patients and the western ones, this retrospective study aims to investigate the incidence of LARS in Chinese patients undergoing laparoscopic LAR, and to explore perioperative risk factors that might be associated with major LARS. Consequent patients undergoing laparoscopic LAR and free from disease recurrence from January 2015 to May 2021 were issued with LARS questionnaire. Incidence of LARS and patient data were collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed as rectal cancer and underwent radical laparoscopic LAR and straight colorectal/coloanal anastomosis (with or without a protective stoma) by a same surgical team

Exclusion Criteria:

either local or distal recurrence, severe complications such as postoperative anastomotic leakage, failure of protective stoma closure, data missed and no responding to LARS questionnaire

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: rectal cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 261 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2021-05 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
incidence of LARS | at least 1 months postoperatively
  incidence of Low Anterior Resection Syndrome
incidence of major LARS | at least 1 months postoperatively
  incidence of major Low Anterior Resection Syndrome

CONTACTS AND LOCATIONS:
Locations (1):
- the Third Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No